CLINICAL TRIAL: NCT01489202
Title: Randomized Comparison of the Effects of PLatinum Chromium Everolimus-eluting Stent vs. cobAlT Chromium Everolimus-eluting Stent on inFlammatOry maRkers and Endothelial daMage - The PLATFORM Trial
Brief Title: Effects of DES Platforms on Markers of Endothelial Damage and Inflammation
Acronym: PLATFORM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 655/2011/D
Record Dates: First submitted 2011-12-06; First posted 2011-12-09 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stent; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- platinum chromium EES (Active Comparator): Patients undergoing PCI with stenting will have implantation of platinum chromium everolimus-eluting stents
  Interventions: Device: platinum chromium everolimus-eluting stent
- cobalt chromium everolimus-eluting stent (Active Comparator): Patients undergoing PCI with stenting will have implantation of cobalt chromium everolimus-eluting stents
  Interventions: Device: cobalt chromium everolimus-eluting stent

INTERVENTIONS:
Device: platinum chromium everolimus-eluting stent — An everolimus-eluting stent with a platinum chromium platform
  Other Names: Promus ElementTM, Boston Scientific Corporation, Natick, MA, USA
  Arms: platinum chromium EES
Device: cobalt chromium everolimus-eluting stent — An everolimus-eluting stent with cobalt chromium platform
  Other Names: Xience VTM, Abbott Laboratories, Abbott Park, IL, USA
  Arms: cobalt chromium everolimus-eluting stent

SUMMARY:
Percutaneous coronary intervention (PCI) with stenting may induce endothelial damage/dysfunction and inflammatory reactions, which in turn delay healing and endothelialization and may lead to restenosis and atherosclerosis within the stented segments. Drugs and polymers are considered the protagonists of these pathophysiologic processes whereas the role of stent platforms remains poorly defined.It remains unknown, conversely, if stent platforms affect the extent of post-PCI endothelial damage and inflammation.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) with stenting may induce endothelial damage/dysfunction and inflammatory reactions, which in turn delay healing and endothelialization and may lead to restenosis and atherosclerosis within the stented segments.

Drugs and polymers are considered the protagonists of these pathophysiologic processes whereas the role of stent platforms remains poorly defined.

Due to advances in stent technology, stent platforms have evolved from the cobalt-chromium (CoCr) to the platinum-chromium (PtCr) stent series. At present, the PROMUS Element stent (which uses the PtCr platform) employs an identical polymer, drug, drug formulation and dose density to the CoCr XIENCE V stent.

The PLATINUM WH trial is the only randomized trial comparing the PROMUS Element stent with the XIENCE V stent in a total of 1,530 patients. The study met its primary end-point demonstrating that the PROMUS Element stent is non-inferior to the XIENCE V stent. The 12-month rare of target lesion failure was 3.4% in the PROMUS Element stent and 2.9% in the XIENCE V stent.

Pre-clinical animal studies, however, suggest that the PtCr platform might have important advantages over the CrCo platform, as improved vascular compatibility and early and late healing for PtCr devices compared with CoCr stents have been demonstrated.

In a rabbit denudation model, it was shown that at 14 days the luminal surface area is incompletely endothelialised with the CrCo stents but nearly complete for the PtCr stents. Similarly, another experimental study has shown that overall strut coverage, including endothelial cell coverage plus non-endothelial cell coverage (focal platelet and fibrin aggregates inter-mixed with red blood cells and inflammatory cells), is significantly lower at 14 days with the CoCr stent than with the PtCr OMEGA stent. Additionally, a recent investigation has shown that the thinner-strut PtCr stent is associated with reduced fibrin deposition and more rapid fibrin clearance in porcine coronary arteries compared with CrCo stent, thus suggesting that the PtCr stent platform may induce less injury compared with previous-generation platforms.

The primary objective of this study is to perform a randomized comparison of the biohumoral effects of platinum chromium everolimus-eluting stent (PtCr EES) vs. cobalt chromium everolimus-eluting stent (CoCr EES), i.e. stents with different platforms but identical drug and polymer.

ELIGIBILITY:
Inclusion Criteria:

* A de novo native coronary artery lesions (reference vessel diameter:2.5-3.75 mm)
* Class I indication to elective percutaneous coronary intervention
* Stable conditions and no recent acute coronary syndromes
* Normal baseline values of markers of myocardial damage (creatine kinase, creatine kinase-MB, myoglobin, and troponin I)
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Post-PCI changes in markers of endothelial damage | Baseline and 24 hours after PCI
  Changes 24 hours after PCI in the following indexes of endothelial damage:
  1. von Willebrand Factor (vWF)
  2. sE-selectin
  3. Vascular cell adhesion molecule (sVCAM-1)
  4. Intercellular adhesion molecule (sICAM-1)
Post-PCI changes in markers of inflammation | Baseline and 24 hours after PCI
  Changes 24 hours after PCI in the following inflammatory markers:
  1. C-reactive protein (CPR)
  2. Fibrinogen
  3. Plasminogen activator inhibitor (PAI-1)
  4. Interleukin-6 (IL-6)

SECONDARY OUTCOMES:
12-month rate of MACE | Up to 12 months
  12-months incidence of major adverse cardiac events (MACE-death, myocardial infarction, target vessel revascularization)

CONTACTS AND LOCATIONS:
Locations (1):
- University La Sapienza, Rome, Italy

REFERENCES:
- [Derived] Pelliccia F, Del Prete G, Del Prete A, Greco C, Gaudio C. Effects of percutaneous coronary intervention and stenting with different drug-eluting coatings and platforms on endothelial damage and inflammation. Int J Cardiol. 2012 Apr 19;156(2):242-3. doi: 10.1016/j.ijcard.2012.01.059. Epub 2012 Feb 22. No abstract available. PMID 22360944